CLINICAL TRIAL: NCT02869802
Title: Prospectively Defining Metastatic Pancreatic Ductal Adenocarcinoma Subtypes by Comprehensive Genomic Analysis
Acronym: PanGen
Status: Recruiting | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Terry Fox Research Institute (Other); BC Cancer Foundation (Other); Pancreas Centre BC (Other); American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: H20-02375; H16-00291 (Other: University of British Columbia)
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Pancreatic Cancer
Keywords: Cancer; Pancreatic Cancer; Advanced Pancreatic Ductal Adenocarcinoma; PDAC; Genomic Analysis; Molecular subtyping
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumour tissue biopsy samples Archival tumour tissue samples Whole blood samples Plasma samples Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Biopsy Cohort: Participants will undergo a tumour biopsy at baseline and an optional tumour biopsy at disease progression.
  Participants will undergo serial collection of plasma and serum samples.
  Interventions: Procedure: Tumour Biopsy; Other: Serial Collection of Plasma and Serum Samples
- Archival Cohort: Genomic analyses will be performed on participants' archival tumour samples.
  Participants will undergo serial collection of plasma and serum samples.
  Interventions: Other: Serial Collection of Plasma and Serum Samples

INTERVENTIONS:
Procedure: Tumour Biopsy — If there is the presence of a tumour lesion amenable to core needle biopsy as judged by a staff interventional radiologist, a minimum of 3 tumour cores will be obtained under CT or US guidance.
  Groups: Biopsy Cohort
Other: Serial Collection of Plasma and Serum Samples — Participants will undergo serial collection of plasma and serum samples at baseline and every cycle of chemotherapy or every 4 weeks, whichever is longer, until end of study.

SUMMARY:
Researchers are looking for better ways of understanding and treating pancreatic cancer. The purpose of this study is to see how useful it is to look for changes and characteristics in your genes (molecules that contain instructions for the development and functioning of the cells) and the genes within the tumour. These characteristics may be useful in choosing treatments for patients in the future. Changes (mutations) in genes have been shown to be an important characteristic in cancers. Looking at differences in genes in patients with advanced pancreatic ductal adenocarcinomas and comparing this information with response to their initial chemotherapy treatment may help to learn which treatments may be better for certain patients after initial treatment.

DETAILED DESCRIPTION:
This is a prospective non-randomized study of patients with metastatic pancreatic ductal adenocarcinoma (PDAC) undergoing first-line systemic chemotherapy with either folinic acid, fluorouracil, irinotecan, and oxaliplatin (FOLFIRINOX) or gemcitabine and nab-paclitaxel (GP)-based regimens, where tumour samples, baseline and serial blood samples, and standardized clinical and radiological assessments will be obtained. Patients planned for treatment with an investigational agent(s) within a clinical trial using either FOLFIRINOX or GP as the chemotherapy backbone will also be eligible, as long other eligibility criteria for the study are met.

A total of 190 patients will be recruited over the study period. Patients will undergo fresh tumour biopsy at study baseline for comprehensive molecular characterization (biopsy cohort). Patients whose biopsy was unable to undergo whole genome and transcriptome sequencing (e.g. due to insufficient tumour content) but fulfill all other eligibility criteria will comprise the archival cohort, where limited genomic analyses will be performed on archival tumour samples. Patients with a radiological diagnosis of metastatic PDAC without a confirmatory histological diagnosis may be eligible; in these cases, tumour biopsy for establishing a pathological diagnosis will be given first priority. Remaining tumour samples will be used for research purposes only after the diagnosis of PDAC has been established. In the rare event (<5%) where the histological diagnosis is other than PDAC, patients will be censored from the study and all tumour materials stored for future clinical use outside of this study.

All patients will undergo serial collection of plasma and serum samples at baseline and every cycle of chemotherapy or every 4 weeks, whichever is longer, until end of study. These samples will be used for exploratory biomarker analyses. Serum cancer antigen 19-9 (CA19-9), also known as carbohydrate antigen 19-9, will also be measured at baseline and every cycle of chemotherapy or every 4 weeks thereafter, whichever is longer, as part of routine standard of care until end of study. In addition, a whole blood sample will be collected at baseline to study germline DNA variants. CT chest, abdomen and pelvis will be performed at baseline and every 8 weeks, with radiological response to therapy assessed using RECIST 1.1.

Patients must have at least one tumour lesion amenable to biopsy from which a minimum of 3 tumour cores can be safely obtainable under CT or ultrasound guidance, as assessed by a staff interventional radiologist. A maximum of 5 tumour cores will be taken from each patient at baseline prior to treatment with FOLFIRINOX or GP. At the time of radiological disease progression, an optional second tumour biopsy will be collected from patients in the biopsy cohort to study changes in the molecular characteristics of tumours under the selection pressure of first-line systemic therapy. This tumour biopsy will be performed using exactly the same procedures described for the baseline biopsy. Tumour biopsies will be coordinated with the British Columbia (BC) Cancer Personalized Oncogenomics (POG) program and the data and/or samples shared between the two studies to avoid re-sampling the patient for both POG and PanGen, if the patient is participating in both studies. Molecular analyses will be performed by BC Cancer. Depending on the amount of tumour material obtained from each patient, molecular analyses will be prioritized to first establish or confirm histological diagnosis and then use for whole genome sequencing, whole transcriptome sequencing, proteomics, and patient-derived models.

The primary endpoint of PanGen is the generation of molecular and phenotypic signatures of individual tumours in a clinically relevant timeframe. The signature data will be correlated with clinical outcome. One of the key strengths of this cohort approach will be the rigorous annotation of PDAC patients' clinical features and outcomes to all treatments (first-line and other) linked to the molecular profile. The investigators have the potential to be nimble as more data is generated, more hypotheses can be explored and others fine-tuned or eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Histological and/or radiological diagnosis of metastatic PDAC. Patients without a histological diagnosis of PDAC must undergo confirmatory tumour biopsy prior to treatment start date.
* Planned for first-line systemic therapy with FOLFIRINOX or GP, either in routine care or in combination with an investigational agent(s) within a clinical trial.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function
* Life expectancy of > 90 days as judged by the investigator
* Ability to give informed consent
* Measurable disease by RECIST 1.1
* Presence of a tumour lesion amenable to core needle biopsy as judged by a staff interventional radiologist. A minimum of 3 tumour cores must be safely obtainable under CT or US guidance.
* Fit enough to safely undergo a tumour biopsy as judged by the investigator
* Ability to lie supine for > 60 minutes

Patients in the archival cohort must also fulfil the following criteria:

* Archival tumour sample available (either a previous tumour diagnostic biopsy or resection specimen)

Exclusion Criteria:

* Absence of distant or lymph node metastases. Patients with borderline resectable or locally advanced PDAC are not eligible.
* Received prior systemic therapy (chemotherapy or any other anti-cancer agent) in the advanced setting. Patients who received adjuvant chemotherapy after surgical resection of early stage disease are eligible.
* Currently receiving anti-cancer therapy (chemotherapy or any other anti-cancer agent)
* Not fit for combination chemotherapy as judged by the investigator
* Presence of brain metastases
* Female patients with positive pregnancy test
* Patients who are not safe to include in the study as judged by the investigator for any medical or non-medical reason
* Unable to comply with study assessments and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic PDAC undergoing first-line systemic therapy with either FOLFIRINOX or GP-based regimens.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2016-10-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of days between biopsy and return of comprehensive genomic results. | An average of 8 weeks
  The primary endpoint is the assessment of the feasibility of returning comprehensive genomic results within a clinically meaningful timeframe. Specifically the primary endpoint is return of genomic data by 8 weeks from the time of biopsy. This endpoint will be met if the analysis data is available within 8 weeks for 80% of the first 50 patients whose tumours are successfully sequenced.

SECONDARY OUTCOMES:
Response Rate | Up to an average of 1 year
  Response rate defined as the percentage of patients with complete (CR) or partial response (PR) per RECIST 1.1
Disease Control Rate | Up to an average of 1 year
  Disease control rate defined as the percentage of patients who experience CR, PR, or stable disease by RECIST 1.1
Duration of Response | Up to an average of 1 year
  Duration of response defined as the interval between the first date of CR or PR and the earliest date of disease progression or death due to any cause
Progression-Free Survival | Up to an average of 1 year
  Progression-free survival (PFS) defined as the interval between the date of registration and the earliest date of disease progression or death due to any cause
Overall Survival | Up to an average of 1 year
  Overall survival (OS) defined as the interval between the date of registration and the date of death.

OTHER OUTCOMES:
Engraftment rate of patient-derived xenografts | 5 years
Success rate of establishing patient-derived organoids | 5 years
DNA damage repair pathways | 5 years
  Percentage of patients with somatic or germline alterations in DNA damage repair pathways
Hypermutated phenotype | 5 years
  Percentage of patients with a hypermutated phenotype
Mismatch repair deficiency | 5 years
  Percentage of patients with mismatch repair deficiency
Neo-antigen load | 5 years
  Percentage of patients with a high tumour neo-antigen load
Targetable mutations | 5 years
  Percentage of patients with rare but targetable mutations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Renouf, MD, Principal Investigator — BC Cancer
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurton S, MacDonald F, Porter G, Walsh M, Molinari M. The current state of pancreatic cancer in Canada: incidence, mortality, and surgical therapy. Pancreas. 2014 Aug;43(6):879-85. doi: 10.1097/MPA.0000000000000147. PMID 24763076
- [Background] Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian Cancer Statistics 2015. Toronto, ON: Canadian Cancer Society; 2015.
- [Background] Sener SF, Fremgen A, Menck HR, Winchester DP. Pancreatic cancer: a report of treatment and survival trends for 100,313 patients diagnosed from 1985-1995, using the National Cancer Database. J Am Coll Surg. 1999 Jul;189(1):1-7. doi: 10.1016/s1072-7515(99)00075-7. PMID 10401733
- [Background] Garcea G, Dennison AR, Pattenden CJ, Neal CP, Sutton CD, Berry DP. Survival following curative resection for pancreatic ductal adenocarcinoma. A systematic review of the literature. JOP. 2008 Mar 8;9(2):99-132. PMID 18326920
- [Background] Rothenberg ML, Moore MJ, Cripps MC, Andersen JS, Portenoy RK, Burris HA 3rd, Green MR, Tarassoff PG, Brown TD, Casper ES, Storniolo AM, Von Hoff DD. A phase II trial of gemcitabine in patients with 5-FU-refractory pancreas cancer. Ann Oncol. 1996 Apr;7(4):347-53. doi: 10.1093/oxfordjournals.annonc.a010600. PMID 8805925
- [Background] Glimelius B, Hoffman K, Sjoden PO, Jacobsson G, Sellstrom H, Enander LK, Linne T, Svensson C. Chemotherapy improves survival and quality of life in advanced pancreatic and biliary cancer. Ann Oncol. 1996 Aug;7(6):593-600. doi: 10.1093/oxfordjournals.annonc.a010676. PMID 8879373
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Mahaseth H, Brutcher E, Kauh J, Hawk N, Kim S, Chen Z, Kooby DA, Maithel SK, Landry J, El-Rayes BF. Modified FOLFIRINOX regimen with improved safety and maintained efficacy in pancreatic adenocarcinoma. Pancreas. 2013 Nov;42(8):1311-5. doi: 10.1097/MPA.0b013e31829e2006. PMID 24152956
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- [Background] Seicean A, Petrusel L, Seicean R. New targeted therapies in pancreatic cancer. World J Gastroenterol. 2015 May 28;21(20):6127-45. doi: 10.3748/wjg.v21.i20.6127. PMID 26034349
- [Background] Collisson EA, Sadanandam A, Olson P, Gibb WJ, Truitt M, Gu S, Cooc J, Weinkle J, Kim GE, Jakkula L, Feiler HS, Ko AH, Olshen AB, Danenberg KL, Tempero MA, Spellman PT, Hanahan D, Gray JW. Subtypes of pancreatic ductal adenocarcinoma and their differing responses to therapy. Nat Med. 2011 Apr;17(4):500-3. doi: 10.1038/nm.2344. Epub 2011 Apr 3. PMID 21460848
- [Background] Biankin AV, Waddell N, Kassahn KS, Gingras MC, Muthuswamy LB, Johns AL, Miller DK, Wilson PJ, Patch AM, Wu J, Chang DK, Cowley MJ, Gardiner BB, Song S, Harliwong I, Idrisoglu S, Nourse C, Nourbakhsh E, Manning S, Wani S, Gongora M, Pajic M, Scarlett CJ, Gill AJ, Pinho AV, Rooman I, Anderson M, Holmes O, Leonard C, Taylor D, Wood S, Xu Q, Nones K, Fink JL, Christ A, Bruxner T, Cloonan N, Kolle G, Newell F, Pinese M, Mead RS, Humphris JL, Kaplan W, Jones MD, Colvin EK, Nagrial AM, Humphrey ES, Chou A, Chin VT, Chantrill LA, Mawson A, Samra JS, Kench JG, Lovell JA, Daly RJ, Merrett ND, Toon C, Epari K, Nguyen NQ, Barbour A, Zeps N; Australian Pancreatic Cancer Genome Initiative; Kakkar N, Zhao F, Wu YQ, Wang M, Muzny DM, Fisher WE, Brunicardi FC, Hodges SE, Reid JG, Drummond J, Chang K, Han Y, Lewis LR, Dinh H, Buhay CJ, Beck T, Timms L, Sam M, Begley K, Brown A, Pai D, Panchal A, Buchner N, De Borja R, Denroche RE, Yung CK, Serra S, Onetto N, Mukhopadhyay D, Tsao MS, Shaw PA, Petersen GM, Gallinger S, Hruban RH, Maitra A, Iacobuzio-Donahue CA, Schulick RD, Wolfgang CL, Morgan RA, Lawlor RT, Capelli P, Corbo V, Scardoni M, Tortora G, Tempero MA, Mann KM, Jenkins NA, Perez-Mancera PA, Adams DJ, Largaespada DA, Wessels LF, Rust AG, Stein LD, Tuveson DA, Copeland NG, Musgrove EA, Scarpa A, Eshleman JR, Hudson TJ, Sutherland RL, Wheeler DA, Pearson JV, McPherson JD, Gibbs RA, Grimmond SM. Pancreatic cancer genomes reveal aberrations in axon guidance pathway genes. Nature. 2012 Nov 15;491(7424):399-405. doi: 10.1038/nature11547. Epub 2012 Oct 24. PMID 23103869
- [Background] Waddell N, Pajic M, Patch AM, Chang DK, Kassahn KS, Bailey P, Johns AL, Miller D, Nones K, Quek K, Quinn MC, Robertson AJ, Fadlullah MZ, Bruxner TJ, Christ AN, Harliwong I, Idrisoglu S, Manning S, Nourse C, Nourbakhsh E, Wani S, Wilson PJ, Markham E, Cloonan N, Anderson MJ, Fink JL, Holmes O, Kazakoff SH, Leonard C, Newell F, Poudel B, Song S, Taylor D, Waddell N, Wood S, Xu Q, Wu J, Pinese M, Cowley MJ, Lee HC, Jones MD, Nagrial AM, Humphris J, Chantrill LA, Chin V, Steinmann AM, Mawson A, Humphrey ES, Colvin EK, Chou A, Scarlett CJ, Pinho AV, Giry-Laterriere M, Rooman I, Samra JS, Kench JG, Pettitt JA, Merrett ND, Toon C, Epari K, Nguyen NQ, Barbour A, Zeps N, Jamieson NB, Graham JS, Niclou SP, Bjerkvig R, Grutzmann R, Aust D, Hruban RH, Maitra A, Iacobuzio-Donahue CA, Wolfgang CL, Morgan RA, Lawlor RT, Corbo V, Bassi C, Falconi M, Zamboni G, Tortora G, Tempero MA; Australian Pancreatic Cancer Genome Initiative; Gill AJ, Eshleman JR, Pilarsky C, Scarpa A, Musgrove EA, Pearson JV, Biankin AV, Grimmond SM. Whole genomes redefine the mutational landscape of pancreatic cancer. Nature. 2015 Feb 26;518(7540):495-501. doi: 10.1038/nature14169. PMID 25719666
- [Background] Moffitt RA, Marayati R, Flate EL, Volmar KE, Loeza SG, Hoadley KA, Rashid NU, Williams LA, Eaton SC, Chung AH, Smyla JK, Anderson JM, Kim HJ, Bentrem DJ, Talamonti MS, Iacobuzio-Donahue CA, Hollingsworth MA, Yeh JJ. Virtual microdissection identifies distinct tumor- and stroma-specific subtypes of pancreatic ductal adenocarcinoma. Nat Genet. 2015 Oct;47(10):1168-78. doi: 10.1038/ng.3398. Epub 2015 Sep 7. PMID 26343385
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Golan T, Kanji ZS, Epelbaum R, Devaud N, Dagan E, Holter S, Aderka D, Paluch-Shimon S, Kaufman B, Gershoni-Baruch R, Hedley D, Moore MJ, Friedman E, Gallinger S. Overall survival and clinical characteristics of pancreatic cancer in BRCA mutation carriers. Br J Cancer. 2014 Sep 9;111(6):1132-8. doi: 10.1038/bjc.2014.418. Epub 2014 Jul 29. PMID 25072261
- [Background] Kaufman B, Shapira-Frommer R, Schmutzler RK, Audeh MW, Friedlander M, Balmana J, Mitchell G, Fried G, Stemmer SM, Hubert A, Rosengarten O, Steiner M, Loman N, Bowen K, Fielding A, Domchek SM. Olaparib monotherapy in patients with advanced cancer and a germline BRCA1/2 mutation. J Clin Oncol. 2015 Jan 20;33(3):244-50. doi: 10.1200/JCO.2014.56.2728. Epub 2014 Nov 3. PMID 25366685
- [Background] Mateo J, Carreira S, Sandhu S, Miranda S, Mossop H, Perez-Lopez R, Nava Rodrigues D, Robinson D, Omlin A, Tunariu N, Boysen G, Porta N, Flohr P, Gillman A, Figueiredo I, Paulding C, Seed G, Jain S, Ralph C, Protheroe A, Hussain S, Jones R, Elliott T, McGovern U, Bianchini D, Goodall J, Zafeiriou Z, Williamson CT, Ferraldeschi R, Riisnaes R, Ebbs B, Fowler G, Roda D, Yuan W, Wu YM, Cao X, Brough R, Pemberton H, A'Hern R, Swain A, Kunju LP, Eeles R, Attard G, Lord CJ, Ashworth A, Rubin MA, Knudsen KE, Feng FY, Chinnaiyan AM, Hall E, de Bono JS. DNA-Repair Defects and Olaparib in Metastatic Prostate Cancer. N Engl J Med. 2015 Oct 29;373(18):1697-708. doi: 10.1056/NEJMoa1506859. PMID 26510020
- [Background] Hahn SA, Greenhalf B, Ellis I, Sina-Frey M, Rieder H, Korte B, Gerdes B, Kress R, Ziegler A, Raeburn JA, Campra D, Grutzmann R, Rehder H, Rothmund M, Schmiegel W, Neoptolemos JP, Bartsch DK. BRCA2 germline mutations in familial pancreatic carcinoma. J Natl Cancer Inst. 2003 Feb 5;95(3):214-21. doi: 10.1093/jnci/95.3.214. PMID 12569143
- [Background] Roberts NJ, Jiao Y, Yu J, Kopelovich L, Petersen GM, Bondy ML, Gallinger S, Schwartz AG, Syngal S, Cote ML, Axilbund J, Schulick R, Ali SZ, Eshleman JR, Velculescu VE, Goggins M, Vogelstein B, Papadopoulos N, Hruban RH, Kinzler KW, Klein AP. ATM mutations in patients with hereditary pancreatic cancer. Cancer Discov. 2012 Jan;2(1):41-6. doi: 10.1158/2159-8290.CD-11-0194. Epub 2011 Dec 29. PMID 22585167
- [Background] Jones S, Hruban RH, Kamiyama M, Borges M, Zhang X, Parsons DW, Lin JC, Palmisano E, Brune K, Jaffee EM, Iacobuzio-Donahue CA, Maitra A, Parmigiani G, Kern SE, Velculescu VE, Kinzler KW, Vogelstein B, Eshleman JR, Goggins M, Klein AP. Exomic sequencing identifies PALB2 as a pancreatic cancer susceptibility gene. Science. 2009 Apr 10;324(5924):217. doi: 10.1126/science.1171202. Epub 2009 Mar 5. PMID 19264984
- [Background] Holter S, Borgida A, Dodd A, Grant R, Semotiuk K, Hedley D, Dhani N, Narod S, Akbari M, Moore M, Gallinger S. Germline BRCA Mutations in a Large Clinic-Based Cohort of Patients With Pancreatic Adenocarcinoma. J Clin Oncol. 2015 Oct 1;33(28):3124-9. doi: 10.1200/JCO.2014.59.7401. Epub 2015 May 4. PMID 25940717
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Riazy M, Kalloger SE, Sheffield BS, Peixoto RD, Li-Chang HH, Scudamore CH, Renouf DJ, Schaeffer DF. Mismatch repair status may predict response to adjuvant chemotherapy in resectable pancreatic ductal adenocarcinoma. Mod Pathol. 2015 Oct;28(10):1383-9. doi: 10.1038/modpathol.2015.89. Epub 2015 Jul 31. PMID 26226846
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Wang J, Chen J, Chang P, LeBlanc A, Li D, Abbruzzesse JL, Frazier ML, Killary AM, Sen S. MicroRNAs in plasma of pancreatic ductal adenocarcinoma patients as novel blood-based biomarkers of disease. Cancer Prev Res (Phila). 2009 Sep;2(9):807-13. doi: 10.1158/1940-6207.CAPR-09-0094. Epub 2009 Sep 1. PMID 19723895
- [Background] Bathe OF, Shaykhutdinov R, Kopciuk K, Weljie AM, McKay A, Sutherland FR, Dixon E, Dunse N, Sotiropoulos D, Vogel HJ. Feasibility of identifying pancreatic cancer based on serum metabolomics. Cancer Epidemiol Biomarkers Prev. 2011 Jan;20(1):140-7. doi: 10.1158/1055-9965.EPI-10-0712. Epub 2010 Nov 23. PMID 21098649
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Background] Wong HL, Zhao EY, Jones MR, Reisle CR, Eirew P, Pleasance E, Grande BM, Karasinska JM, Kalloger SE, Lim HJ, Shen Y, Yip S, Morin RD, Laskin J, Marra MA, Jones SJM, Schrader KA, Schaeffer DF, Renouf DJ. Temporal Dynamics of Genomic Alterations in a BRCA1 Germline-Mutated Pancreatic Cancer With Low Genomic Instability Burden but Exceptional Response to Fluorouracil, Oxaliplatin, Leucovorin, and Irinotecan. JCO Precis Oncol. 2018 Oct 19;2:PO.18.00057. doi: 10.1200/PO.18.00057. eCollection 2018. No abstract available. PMID 32913994
- [Background] Jones MR, Williamson LM, Topham JT, Lee MKC, Goytain A, Ho J, Denroche RE, Jang G, Pleasance E, Shen Y, Karasinska JM, McGhie JP, Gill S, Lim HJ, Moore MJ, Wong HL, Ng T, Yip S, Zhang W, Sadeghi S, Reisle C, Mungall AJ, Mungall KL, Moore RA, Ma Y, Knox JJ, Gallinger S, Laskin J, Marra MA, Schaeffer DF, Jones SJM, Renouf DJ. NRG1 Gene Fusions Are Recurrent, Clinically Actionable Gene Rearrangements in KRAS Wild-Type Pancreatic Ductal Adenocarcinoma. Clin Cancer Res. 2019 Aug 1;25(15):4674-4681. doi: 10.1158/1078-0432.CCR-19-0191. Epub 2019 May 8. PMID 31068372
- [Background] Heining C, Horak P, Uhrig S, Codo PL, Klink B, Hutter B, Frohlich M, Bonekamp D, Richter D, Steiger K, Penzel R, Endris V, Ehrenberg KR, Frank S, Kleinheinz K, Toprak UH, Schlesner M, Mandal R, Schulz L, Lambertz H, Fetscher S, Bitzer M, Malek NP, Horger M, Giese NA, Strobel O, Hackert T, Springfeld C, Feuerbach L, Bergmann F, Schrock E, von Kalle C, Weichert W, Scholl C, Ball CR, Stenzinger A, Brors B, Frohling S, Glimm H. NRG1 Fusions in KRAS Wild-Type Pancreatic Cancer. Cancer Discov. 2018 Sep;8(9):1087-1095. doi: 10.1158/2159-8290.CD-18-0036. Epub 2018 May 25. PMID 29802158
- [Background] Beg MS, Gupta A, Sher D, Ali S, Khan S, Gao A, Stewart T, Ahn C, Berry J, Mortensen EM. Impact of Concurrent Medication Use on Pancreatic Cancer Survival-SEER-Medicare Analysis. Am J Clin Oncol. 2018 Aug;41(8):766-771. doi: 10.1097/COC.0000000000000359. PMID 28079594
- [Derived] Karasinska JM, Topham JT, Kalloger SE, Jang GH, Denroche RE, Culibrk L, Williamson LM, Wong HL, Lee MKC, O'Kane GM, Moore RA, Mungall AJ, Moore MJ, Warren C, Metcalfe A, Notta F, Knox JJ, Gallinger S, Laskin J, Marra MA, Jones SJM, Renouf DJ, Schaeffer DF. Altered Gene Expression along the Glycolysis-Cholesterol Synthesis Axis Is Associated with Outcome in Pancreatic Cancer. Clin Cancer Res. 2020 Jan 1;26(1):135-146. doi: 10.1158/1078-0432.CCR-19-1543. Epub 2019 Sep 3. PMID 31481506
- See also: Integrated Addendum to International Council for Harmonization (ICH) E6(R1): Guideline for Good Clinical Practice ICH E6(R2) — https://database.ich.org/sites/default/files/E6_R2_Addendum.pdf